## Official Title:

Dealing With Intrusive Thoughts in OCD - a Comparison of Detached Mindfulness and Cognitive Restructuring

## Date of Document:

July12<sup>th</sup>, 2018

## NCT number:

NCT03002753

Data were analyzed using the R package ez (Lawrence, 2016) and IBM SPSS Statistics (SPSS) 25.0. Comparability of groups at baseline was analyzed by calculating independent t-tests for continuous variables and  $\chi^2$ -test for categorical variables. In order to evaluate the efficacy of treatments, a 2x2x2 mixed ANOVA was run with the within-subjects factor time, referring to the various assessment points, and the between-subjects factors waitlist (WL/NWL) and treatment condition (CT/MCT). In contrast to the calculation of effect sizes described below this ANOVA excluded the Post assessment data from subjects in the waitlist group towards a conservative testing procedure, so that the definition of time points differed between WL and NWL groups: In both groups, TI referred to Pre1 data, however, T2 referred to Pre2 data in the WL group and to Post data in the NWL, thus separating effects of time and treatment separately. The use of the R package ez involved the computation of the generalized eta squared statistic ( $\eta_G^2$ ) in order to display the amount of explained variance (Olejnik & Algina, 2003).

The calculation of effect sizes (Cohen's d) was based on the whole data set including the Post data from WL subjects, which was based on the a priori assumption of *time* not exhibiting a main effect. Due to this assumption, Pre2 data were not used in the calculation of effect sizes. Three effect sizes (Pre1-Post, Post-FU, and Pre1-FU) were calculated for each treatment condition as follows, using pooled standard deviations ( $SD_{Pre1}$ : 3.385;  $SD_{Post}$ : 5.789) instead of separate standard deviations for CT and MCT (x = mean Y-BOCS score, SD = standard deviation):  $d_1 = \frac{x_{Pre1} - x_{Post}}{SD_{Pre1}}$ ,  $d_2 = \frac{x_{Post} - x_{FU}}{SD_{Post}}$ ,  $d_3 = \frac{x_{Pre1} - x_{FU}}{SD_{Pre1}}$ .

Moreover, in order to display the *amount* of improvement, clinically significant change was assessed as proposed by Jacobson & Truax (1991). It was defined by a combination of two criteria: (1) *reliable improvement*:  $RC = \frac{x_2 - x_1}{S_{diff}}$ , with  $x_1$  representing a person's Y-BOCS score at Pre1 assessment,  $x_2$  referring to a person's Y-BOCS score at Post

assessment, and  $S_{diff}$  denoting being the standard error of difference scores (based on the internal consistency of the German version of the Y-BOCS (r = .80, ) as reported by Jacobsen, Kloss, Fricke, Hand, and Moritz (2003). Based on our calculations, a decrease of 5 points or more on the Y-BOCS indicated was used as an index of reliable improvement. (2) recovery criterion:  $a = M_1 - 2*SD_1$ , with  $M_1$  representing the mean Y-BOCS score of the sample at Pre1 assessment and SD<sub>1</sub> referring to the corresponding standard deviation. A post assessment Y-BOCS score of a = 17.9 or less indicated recovery. A reliable change was presumed if participants displayed a post-assessment Y-BOCS score of 17.9 or less (recovery criterion) and a minimal Pre1-Post change of 5 -points on the Y-BOCS (reliable improvement criterion).